CLINICAL TRIAL: NCT00153283
Title: Randomised, Placebo Controlled, Double Blind, Parallel Group 3-Months Study of Gabapentin Efficacy in Asthma Therapy
Brief Title: Study of Efficacy of Gabapentin in Therapy of Bronchial Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre of Chinese Medicine, Georgia (Other)
Collaborators: Rea Rehabilitation Centre, Georgia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTP-0904-GP-0404
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Bronchial Asthma
Keywords: Bronchial asthma; Gabapentin; Antiepileptic drug; Efficacy
MeSH Terms: conditions — Asthma | interventions — Gabapentin

INTERVENTIONS:
Drug: Gabapentin

SUMMARY:
The purpose of this study is to determine whether antiepileptic drug gabapentin is effective in the treatment of chronic asthma.

DETAILED DESCRIPTION:
Effective therapy of asthma still remains quite serious problem. According GINA definition, asthma is an inflammatory disorder. Consequently, modern pharmacotherapy of asthma provides wide use of anti-inflammatory drugs. But asthma also is a paroxysmal disorder: many specialists and even some guidelines underline paroxysmal clinical picture of asthma. Besides this, according to some authors, neurogenic inflammation may play important role in asthma mechanism. But some other neurogenic inflammatory paroxysmal disorders exist, and they are migraine and trigeminal neuralgia. Some antiepileptic drugs, like carbamazepine and valproate, are very effective in therapy of migraine and trigeminal neuralgia - more than in 80% of cases. If bronchial asthma also is paroxysmal inflammatory disease, like migraine and trigeminal neuralgia, it is possible that some antiepileptic drugs also are very effective in asthma therapy.

We performed a double-blind, placebo-controlled 3-month trial for evaluation of gabapentin efficacy in therapy of bronchial asthma. Gabapentin is antiepileptic drug of new generation, produced by Pfizer.

Comparison: Patients received investigational drug in addition to their usual routine antiasthmatic treatment, compared to patients received placebo in addition to their usual routine antiasthmatic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have given their informed consent before commencing the procedures specified in the protocol, indicating that they understand the objectives of the study and are willing to adhere to the procedures described in the protocol.
* Males or females.
* Patient aged between 16 and 65 years.
* Out patients.
* Non smokers or ex-smokers, having stopped smoking > 1 year.
* Patients with an established (i.e. at least one year) clinical history of asthma.
* Absence of long-term remissions of asthma (lasting more than 1 month)
* Poorly controlled asthma, due to various reasons.
* Patients with a FEV1 reversibility of at least 12% from initial level after 400 mcg salbutamol inhalation (4 puffs of salbutamol MDI, 100 mcg per puff). Patients whose FEV1 reversibility was 12% within the past 12 months are acceptable, providing that the records are available to the investigator.
* Patients able to swallow capsules, able to understand and complete diary cards and to record their PEFR using a peak-flow meter.

Exclusion Criteria:

* Long-term history of smoking (3 years and more)
* History or presence of cardiovascular, renal, neurologic, psychiatric, liver, immunologic, endocrine, infection or other diseases or dysfunctions if they are clinically significant. A clinically significant disease is defined as one which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
* Patients with a recent history (< 1 year) of myocardial infarction and/or (< 3 years) of heart failure or patients with any cardiac arrhythmia requiring drug therapy.
* History of cancer within the past 5 years.
* Patients with active tuberculosis with indication for treatment.
* Patients with a history of cystic fibrosis, bronchiectasis, chronic bronchitis or emphysema.
* Patients with clinically significant abnormal baseline haematology, blood chemistry or urinalysis or if the abnormal defines a disease listed as an exclusion criterion.
* Patients with known allergy, side effects, intolerance/hypersensitivity to investigational drug
* Patients currently using MAO inhibitors, tricyclic antidepressants, antiepileptic drugs, narcotic agents.
* Pregnant or nursing women and sexually active women with childbearing potential not using a medically approved method of contraception.
* Patients unlikely, unable or unwilling to comply with the requirements of the protocol.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68
Dates: Start 2003-09; Study Completion 2004-04

PRIMARY OUTCOMES:
At 3 months of treatment: Change from baseline of the FEV1 and PEFR (also %predicted); Number of patients without asthma symptoms

SECONDARY OUTCOMES:
At 3 months of treatment: FEV1 before and after salbutamol inhalation; Difference in PEF pm-am (in %); The daily (daytime and night-time) symptoms scores; % of symptom free days during the treatment period; Use of other antiasthmatic medication

CONTACTS AND LOCATIONS:
Overall Officials: Merab Lomia, MD, Principal Investigator — "Rea" Rehabilitation Centre; Tamara Tchelidze, MD, Study Director — CRO Evidence; Manana Tchaia, MD, Study Chair — Centre of Chinese Medicine

REFERENCES:
- See also: Website of Neuroasthma Group — http://www.asthma.ge
- See also: Bronchial asthma as neurogenic paroxysmal inflammatory disease: a randomized trial with carbamazepine — http://www.ncbi.nlm.nih.gov/pubmed/16597501?ordinalpos=2&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum